CLINICAL TRIAL: NCT00000248
Title: Dose Response Trial of Pergolide for Cocaine Dependence
Brief Title: Dose Response Trial of Pergolide for Cocaine Dependence - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-08355-1; R01DA008355 (NIH); R01-08355-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 1997-05

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Pergolide

INTERVENTIONS:
Drug: Pergolide

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of pergolide for treatment of cocaine dependence.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-02

PRIMARY OUTCOMES:
Side effects
Drug use
Retention
Cocaine withdrawal
Compliance
Effectiveness of medication for global improvements

CONTACTS AND LOCATIONS:
Overall Officials: Robert Malcolm, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Malcolm R, Moore JW, Kajdasz DK, Cochrane CE. Pergolide mesylate. Adverse events occurring in the treatment of cocaine dependence. Am J Addict. 1997 Spring;6(2):117-23. doi: 10.3109/10550499709137022. PMID 9134073